CLINICAL TRIAL: NCT02139787
Title: Somali, Latino & Hmong Radio Stories About Children's Healthy Eating and Exercise: A SoLaHmo Pilot Study
Brief Title: Radio Stories About Children's Healthy Eating and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: West Side Community Health Services (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1209S19821-2
Record Dates: First submitted 2014-05-05; First posted 2014-05-15 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension, obesity; Dietary behaviors; Physical activity behaviors; Radio story, entertainment health education; Immigrants; Somali, Latino, Hmong; Families with 3-18 year old children
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radio Story (Experimental): Participants listen to a radio story about a family's' success with preventing or managing hypertension or obesity through diet and physical activity; the focus was for the entire family to implement healthful lifestyle behaviors so the children can learn as well.
  Interventions: Other: Radio Story
- Control -listened to a brochure (Active Comparator): Participants received an audio version of a standard brochure about hypertension or obesity prevention.
  Interventions: Other: Control -listened to a brochure

INTERVENTIONS:
Other: Radio Story
  Arms: Radio Story
Other: Control -listened to a brochure
  Arms: Control -listened to a brochure

SUMMARY:
The purpose of this study is to use a community based participatory action research (CBPAR) approach to 1) create "radio stories" about Somali, Latino and Hmong families' real success stories with hypertension and obesity in managing their disease through implementation of healthful lifestyle behaviors (nutrition and physical activity), and 2) test the effectiveness and acceptability of radio stories on participant intentions to engage in or improve healthful lifestyle behaviors to prevent these disease. Participants in the Intervention condition listened to the "radio stories" and the participants in the control condition listened to an audio brochure with relevant health information. We hypothesized that the intervention participants would report higher intentions to engage in various healthful lifestyle behaviors than the control participants after both participants listened to their respective health information.

DETAILED DESCRIPTION:
Given the high rate of hypertension and obesity in minority and immigrant communities, implementing culturally and linguistically appropriate health promotion activities that improve families' diet and physical activity behaviors is imperative. "Radio Stories" is an education entertainment strategy that has significant potential as a health promotion tool. Through a CBPAR process, we aimed to create and test the effectiveness and acceptability of "SoLaHmo Radio Stories" about changing knowledge and behaviors to prevent or manage hypertension and obesity for Somali, Latino, and Hmong families with children.

Methods: SoLaHmo community researchers interviewed 7 families (3 Somali, 2 Latino, and 2 Hmong) who have successfully implemented lifestyle changes to prevent or manage hypertension or obesity, and then create 6 "radio stories" (2 per ethnic community) based on the families' experiences. To test the stories, we are conducting a two-arm trial that includes 146 participants (obesity: 68, hypertension: 78; 44 Hmong, 49 Latino, and 53 Somali participants). Effectiveness and acceptability of the program will be tested with pre-and post questionnaires.

Anticipated Results: Higher rates of satisfaction, increased knowledge, and increased intention to change healthful lifestyle behaviors in participants receiving the radio stories, as compared to control group participants, will indicate radio story program effectiveness and acceptability.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Key Family Informant Interviews:

* Family self-identifies as Somali, Latino or Hmong
* Family has at least one child between the ages of 3-18 years old
* English or Spanish or Somali or Hmong speaking
* Family identified as having a compelling story with hypertension or obesity

Inclusion Criteria for Intervention and Control Group Participants:

* Self-identified member of Somali, Latino or Hmong communities
* Adult age 18 years and older
* English or Spanish or Somali or Hmong-speaking
* Parent/caregiver is involved with raising children between the ages of 3-18 years

Exclusion Criteria for Key Family Informant Interviews:

* Family does not self-identify as Somali, Latino or Hmong
* Family does not have children between the ages of 3-18 years
* Not English or Spanish or Somali or Hmong speaking
* Parent/caregiver Is not involved with raising children between the ages of 3-18 years

Exclusion criteria for Intervention and Control Group Participants:

* Participants do not self-identify as Somali, Latino or Hmong
* Participants are younger than 18 years
* Participants are not caregivers of children between the ages of 3-18 years
* Not English or Spanish or Somali or Hmong speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Acceptability and effectiveness of radio stories, a health communication intervention that addresses family eating behaviors and physical activity among immigrant Somali, Latino, and Hmong families. | 'From baseline to flow-up which is after listening to radio story or audio brochure - An average of 25 minutes'
  The baseline and follow-up survey questions to test the "radio stories" included 15 items referring to intentions to change or improve a specific diet, physical activity, and health related behavior. There were four Likert scale response categories, from 'strongly disagree' to 'strongly agree.' In addition, the follow-up survey included questions to assess participant perceptions of the radio stories relating to their emotional connection to the story, relevance with their own experience, believability, and increase awareness and concern about hypertension and obesity. In the baseline survey they were questions pertaining to demographics and dietary and physical activity behaviors.

SECONDARY OUTCOMES:
Concern about hypertension and obesity | Baseline and follow-up (immediately after listening to the health information)

CONTACTS AND LOCATIONS:
Overall Officials: Chrisa Arcan, PhD, MHS, MBA, RD, Principal Investigator — Medical School, University of Minnesota
Locations (1):
- West Side Clinic and Community, Saint Paul, Minnesota, United States